CLINICAL TRIAL: NCT06461078
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Effects of Food on the Pharmacokinetics and Safety of Orally Administered Radotinib in Healthy Adults
Brief Title: Clinical Trial to Investigate the Effects of Food on the Pharmacokinetics and Safety of Orally Administered Radotinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RT51KR-PK01
Record Dates: First submitted 2024-05-29; First posted 2024-06-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-06

CONDITIONS: Drug Kinetics

STUDY DESIGN:
Intervention Model Description: Randomized, Open-label, Single-dose, Two-way Crossover
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Treatment Group (Active Comparator): Radotinib 200mg, 2 Tablets, Fasting, Single dose
  Interventions: Drug: Radotinib HCl
- Active Comparator: Control Group (Active Comparator): Radotinib 200mg, 2 Tablets, Standard diet, Single dose
  Interventions: Drug: Radotinib HCl

INTERVENTIONS:
Drug: Radotinib HCl — 1. Brand name/manufacturer: Supect Cap./IL-YANG PHARM. Co., Ltd.
  2. Active ingredient: radotinib HCl 106.8mg (100mg as radotinib) or HCl 213.6mg (200mg as radotinib)
  3. Appearance and formulation: hard capsule with a light blue cap and a body containing pale yellow powder
  4. Storage conditions: Store in an airtight light proof container at room temperature.
  Other Names: SUPECT

SUMMARY:
A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Effects of Food on the Pharmacokinetics and Safety of Orally Administered Radotinib in Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 or older and 55 or younger at the time of screening tests.
2. Men weigh more than 55 kg and women weigh more than 50 kg.
3. Those who have a body mass index of 18.5 kg/m2 or more and less than 27.0 kg/m2.

   ※ Body mass index (body mass index, kg/m2) = Weight (kg)/[Height (m)]2
4. If participants are a woman, participants must apply to one of the following.

   * Menopause (no natural menstruation for at least 2 years)
   * Surgical infertility (hysterectomy or bilateral oophorectomy, tubal ligation, or other infertility)
5. If a male has sex with a female of childbearing age, he/she must agree to use contraception* until at least 28 days after the clinical trial period and the final administration of the clinical trial drug and not to donate sperm.

   *Contraception: Use a combination of vasectomy, intrauterine device, tubal ligation and blocking contraception (male condom, female condom, cervical cap, contraceptive septum, sponge, etc.) or use a combination of two or more blocking contraception when using a biocidal agent.
6. A subject who has fully understood and received sufficient explanation of this clinical trial and has voluntarily decided to participate and agreed in writing to comply with the precautions.

Exclusion Criteria:

1. A person with a history of clinically significant hepatobiliary system (severe hepatic disorder, hyperbilirubinemia, pancreatitis, etc.), kidney (severe renal disorder, acute renal failure, etc.), urethral disorder, nervous system, immune system, respiratory system, endocrine system, cardiovascular system (myocardial infarction, congestive heart failure, unstable angina, bradycardia, long QT syndrome, torsade de points, etc.), blood, tumor, urinary system, psychiatric disorder, or medical history.
2. Those with a history of gastrointestinal diseases (Crohn's disease, ulcerative colitis, etc.) or surgery (except for simple appendectomy or hernia surgery) that can affect the absorption of drugs.
3. A person who has a history of clinically significant hypersensitivity reactions or allergies to drugs or additives (Yellow 5, Sunset Yellow FCF), including ingredients (Radotinib) of clinical trial drugs.
4. A person who was judged to be inappropriate as a test subject in a screening test conducted within 28 days prior to administration of a clinical drug (examination, blood pressure, 12-lead electrocardiogram, physical examination, clinical laboratory examination, etc.).

   * In the case of > 1.5 times the upper limit of AST and ALT normal range in the blood
   * In the case of > 1.5 times the upper limit of Total bilirubin normal range in the blood
   * Estimated Global Film Rate (eGFR) <60 mL/min/1.73 m2 using the Modification of Diet in Regular Disease (MDRD) formula
   * Serum test (hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test) result are positive factors
   * QTcF > 480 msec on electrocardiogram
   * After resting for at least 5 minutes, those who showed a value corresponding to systolic blood pressure>150 mmHg or <90 mmHg, diastolic blood pressure>100 mmHg or <50 mmHg in the vital signs measured at the seat
5. A person who shows suspected symptoms of acute illness (chilliness, fever, diarrhea, stomatitis, redness, infectious symptoms, etc.) at the time of screening tests.
6. A person who has a history of drug abuse or has tested positive in a urine drug screening test within one year of screening.
7. If the tester determines that the following drugs, excluding topical drugs without significant systemic absorption, may affect this test or affect the safety of the test subject within the relevant period.

   * In the case of taking general medicines including health foods and vitamin preparations within 7 days prior to the first administration of clinical trial drugs
   * In the case of taking a prescription drug or herbal medicine within 14 days prior to the first administration date of the clinical trial drug
   * A person who has administered a CYP3A4 inhibitor (ketoconazole, itraconazole, erythromycin, clarithromycin, etc.) or a CYP3A4 inhibitor (dexamethasone, phenytoin, carbamazepine, rifampicin, phenobarbital, St. John's short [hypericum perforatum], etc.) within 30 days prior to the first administration of clinical trial drug
   * A person who has administered antiarrhythmic drugs (amiodarone, disopyramid, propofol, quinidine, totalol, etc.) or other drugs that can extend the QT interval (chloroquine, halofantrine, clarithromycin, haloperidol, methadone, moxifloxacin, bepridil, pimozide, etc.) within 30 days prior to the first administration of clinical trial drug
   * A person who has received a P-glycoprotein derivative such as ritonavir within 30 days prior to the first day of administration of a clinical trial drug
8. A person who has consumed grapefruit-containing food within 7 days prior to the first administration date of clinical trial drugs or cannot be prohibited from taking it during the clinical trial period.
9. A person who continuously smoked excessively or consumed caffeine or alcohol (caffeine: >5 cups/day, alcohol: >210 g/week, tobacco: >10 g/day) or who cannot stop smoking, caffeine and alcohol consumption during each hospitalization period.
10. A person who participated in another clinical trial (including a bioequivalence test) within 180 days prior to the first administration date of the clinical trial drug and received the clinical trial drug (in the case of biological agents, it may be based on an extended period considering a half-life).
11. A person who donated whole blood within 60 days prior to the first administration date of clinical trial drugs or donated component blood within 30 days.
12. A person who received a blood transfusion within 30 days prior to the first administration date of the clinical trial drug.
13. Pregnant or lactating female at the time of screening tests.
14. A person who determines that the tester is inappropriate to participate in clinical trials due to other reasons.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Cmax(Maximum concentration of drug in plasma) | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours
AUClast(Area under the plasma drug concentration-time curve to last concentration) of Radotinib | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours

SECONDARY OUTCOMES:
AUCinf(Area under the plasma drug concentration-time curve from 0 to infinity) of Radotinib | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours
Tmax(Time to maximum plasma concentration) of Radotinib | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours
t1/2(Terminal elimination half-life) of Radotinib | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours
Vd/F(Apparent volume of distribution), CL/F(Apparent clearance) of Radotinib | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours
Cmax of Radotinib metabolites(M1, M2) | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours
Tmaxof Radotinib metabolites(M1, M2) | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours
t1/2, metabolic ratio(AUClast of metabolite/AUClast of Radotinib) of Radotinib metabolites(M1, M2) | Pre-dose(0 hour), after dose 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 32 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours

CONTACTS AND LOCATIONS:
Overall Officials: Minsoo Park, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea